CLINICAL TRIAL: NCT02969642
Title: A Single-center, Sham-controlled, Single Attack Study of Laser Therapy to the Sphenopalatine Ganglion (SPG) in the Acute Treatment of Migraine
Brief Title: Study of Low-level Laser Therapy in the Acute Treatment of Migraine
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The San Francisco Clinical Research Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AP 1001
Record Dates: First submitted 2016-10-20; First posted 2016-11-21 (Estimated); Last update posted 2016-12-02 (Estimated); Status verified 2016-12

CONDITIONS: Migraine Headache
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sham (Sham Comparator): Sham low energy laser using approximately 1/1000 th energy of treatment laser.
  Interventions: Device: Argus Migraine Treatment device
- Treatment (Active Comparator): Treatment laser.
  Interventions: Device: Argus Migraine Treatment device

INTERVENTIONS:
Device: Argus Migraine Treatment device — treatment of Migraines targeting Sphenopalatine ganglion
  Other Names: low energy laser therapy

SUMMARY:
This study evaluates the treatment of migraine pain using low energy laser light to quench migraine signals issuing from the sphenopalatine ganglion (SPG).

DETAILED DESCRIPTION:
This is a double blinded, two arm study, comprising a sham laser and a treatment laser. The sham laser emits approximately 1/1000 the energy of the treatment laser.

It is presumed that pain relief from the treatment laser is achieved by exhausting the release of neurotransmitters from the SPG following laser stimulation. Subjects will be treated and subsequently queried at time intervals for their self-assessment of pain score (VAS). The time intervals include queries at 5 minutes through 2 hours post treatment. Subjects will be further contacted 24 hours and one month post treatment. Adverse events will be monitored and recorded.

ELIGIBILITY:
Inclusion Criteria

* male or female
* aged 18 or older;
* subject diagnosed with migraine according to The International Classification of Headache Disorders- Version 3;
* 1-20 headache days per month;
* history of at least moderate pain if migraine left untreated.

Exclusion Criteria:

* headache on greater than 25 days/month on average for preceding 3 months;
* headache on greater than 25 days in present month;
* headache attributed to: head or neck trauma, cluster headache, specific migraine variants such as basilar artery, ophthalmoplegic, hemiplegic, etc;
* women of child bearing age not using acceptable method of contraception;
* pregnant or nursing women;
* history of malignancy of any organ
* uncontrolled: hypertension, severe psychiatric disorders, or known use of narcotics, analgesic or alcohol abuse;
* light sensitivity;
* retinal disease;
* intranasal pathology.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2016-03; Primary Completion 2017-05 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
Differences between treatment groups in pain free rates at 2 hours post treatment. | 2 hours post treatment

CONTACTS AND LOCATIONS:
Locations (1):
- San Francisco Clinical Research Center, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No